CLINICAL TRIAL: NCT06656975
Title: Social Prescribing and Relationship Cognitive Strategies (SPARCS)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Paul Pfeiffer, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00258121; 5R34MH132808-02 (NIH)
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Social Isolation; Suicidal Ideation
Keywords: Collaborative Care Management; Social Prescribing; Relationship Cognitive Strategies
MeSH Terms: conditions — Social Isolation; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 1 of 3 arms in a 1:1:1 ratio (see Protocol for detailed descriptions).
Who Masked: Outcomes Assessor
Masking Description: To the extent possible, the assessor will be blinded. The study team will track any instances where an assessor becomes unblinded to a participant's arm assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care control group (Other): Participants will receive an informational booklet on improving loneliness and may initiate or continue Collaborative Care for other conditions on a not research basis.
  Besides the baseline survey participants will also take 2 more surveys, 3-months and 6-months from the first survey. Those surveys will ask similar questions and will take about 45 minutes to complete. These can be done online or over the phone with a researcher that will not know the treatment arm assignment.
  Interventions: Other: Enhanced Usual Care
- Brief Cognitive Therapy then Social Prescribing (Experimental): Besides the baseline survey participants will also take 2 more surveys, 3-months and 6-months from the first survey. Those surveys will ask similar questions and will take about 45 minutes to complete. These can be done online or over the phone with a researcher that will not know the treatment arm assignment.
  Interventions: Behavioral: Brief Cognitive Therapy; Behavioral: Social Prescribing
- Social Prescribing then Brief Cognitive Therapy (Experimental): Besides the baseline survey participants will also take 2 more surveys, 3-months and 6-months from the first survey. Those surveys will ask similar questions and will take about 45 minutes to complete. These can be done online or over the phone with a researcher that will not know the treatment arm assignment.
  Interventions: Behavioral: Brief Cognitive Therapy; Behavioral: Social Prescribing

INTERVENTIONS:
Behavioral: Brief Cognitive Therapy — This intervention will be delivered by participants Behavioral Health Care Manager during Collaborative Care Management appointments. These appointments typically take place over video call (telehealth). Each intervention consists of 4 sessions (approximately 20 minutes each), delivered over 3 months. Participants will also receive a one-time introductory session before starting the first intervention. Between sessions, there will be "homework" tasks, such as filling out worksheets or completing goals that are set with the provider.
  The therapy portion of the appointment only will be audio recorded using a voice recorder or secure meeting software. Audio recordings will be reviewed by study staff for training and compliance purposes.
  Arms: Brief Cognitive Therapy then Social Prescribing; Social Prescribing then Brief Cognitive Therapy
Behavioral: Social Prescribing — This intervention will be delivered by participants Behavioral Health Care Manager during Collaborative Care Management appointments. These appointments typically take place over video call (telehealth). Each intervention consists of 4 sessions (approximately 20 minutes each), delivered over 3 months. Participants will also receive a one-time introductory session before starting the first intervention. Between sessions, there will be "homework" tasks, such as filling out worksheets or completing goals that are set with the provider.
  The therapy portion of the appointment only will be audio recorded using a voice recorder or secure meeting software. Audio recordings will be reviewed by study staff for training and compliance purposes.
  Arms: Brief Cognitive Therapy then Social Prescribing; Social Prescribing then Brief Cognitive Therapy
Other: Enhanced Usual Care — Participants will receive an informational booklet on improving loneliness. Participants may initiate or continue Collaborative Care for other conditions on a not research basis.
  Arms: Enhanced Usual Care control group

SUMMARY:
The study team is testing the acceptability and feasibility of two treatments for improving loneliness: Social Prescribing and Brief Cognitive Therapy.

For this pilot study, the study team have adapted these treatments for Collaborative Care and are studying whether these are practical and well-received by patients that might use them.

DETAILED DESCRIPTION:
The study will take place at 2 University of Michigan sites.

ELIGIBILITY:
Inclusion Criteria:

* Screen positive for either or both of the following during routine clinic screening:

  * Social isolation in the past 6 months, according to the screening question "How often do you feel isolated from others?"
  * Suicidal ideation in the past 12 months, according to the 9th item of the Patient Health Questionnaire (HQ-9) (per protocol)
* Loneliness, according to the 3-item version of the University of California, Los Angeles (UCLA) Loneliness Scale (per protocol)
* Are currently receiving or are able to initiate Collaborative Care Management at to participant's study site

Exclusion Criteria:

* Currently receiving or have an active referral for specialty mental health or substance use disorder treatment outside of primary care
* Neurocognitively impaired according to chart diagnosis, self-report on the Eligibility Screening Survey, or inability to answer comprehension check questions during the Informed Consent process (per protocol)
* Unable to participate in the interventions and research assessments due to planned travel or limited phone access (e.g., does not own phone)
* Terminally ill or receiving of palliative care with less than 6 months life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adapted Client Satisfaction Questionnaire - Intervention arms only | 3 and 6 months
  This is an 8-item self-report survey which assesses participant satisfaction with services received.
  SCORING: Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Intervention Helpfulness - Intervention Arms Only | 6 months
  This is a 9-item, self-report study-specific questionnaire that assesses how much participants were helped by the combined study interventions on various cognitive and behavioral factors that impact loneliness. Questions use a 6-point Likert scale where 0 = "Not applicable/Did not work on this" and 6 = "Made things a lot better." SCORING: Scores will range from 0 to 45, with higher scores indicating greater helpfulness.
UCLA Loneliness Scale | Baseline, 3 and 6 months
  This consists of 20 items using 4-point Likert-type response anchors from never feel this way (0) - often feel this way (3) (9 items are reverse coded) for a score range from 10 to 80.
Computer Adaptive Testing - Suicide Scale (CAT-SS) | Baseline, 3 and 6 months
  The CAT-SS is based on multidimensional item response theory (MIRT). Within computer adaptive testing, an individuals' initial item responses are used to determine a provisional estimate of their standing on the measured trait to be used for subsequent item selection. MIRT weighs more severe items more heavily than less severe items in deriving a test score, and provides an estimate of uncertainty that can be used to assess the significance of change for an individual. The measure adaptively selects an average of 10 items per administration from a large bank of approximately 1,000 items. Instead of fixing the items and allowing the precision of measurement to vary, this measure fixes the precision of measurement and allow the items to vary. As a result, measurement is more precise and less burdensome compared with fixed-item standardized measures of suicidal ideation.
Feasibility will be measured by the recruitment goal of 60 participants | 15 months (recruitment period)
Feasibility will be measured by completion rates of follow-up assessments at 3 and 6 months | 3 and 6 months
  The target for this goal = 75%.

SECONDARY OUTCOMES:
Beck Scale for Suicidal Ideation (BSS) | Baseline, 12 and 24 weeks
  The Beck Scale for Suicidal Ideation (BSS) is a self-report 21-item scale that assesses thoughts, plans and intent to commit suicide. All items are rated on a three-point scale (0 to 2). Total scores could range from 0 to 42. No specific cut-off scores exist to classify severity. Higher scores reflect greater suicide risk.
Interpersonal Needs Questionnaire (INQ) | Baseline, 12 and 24 weeks
  This is a 15-item questionnaire that participants answer from not at all (1) to very true (7).
  There is a score range from 15-105 with a higher score indicating higher perceived burdensomeness.
  There are 6 items that are reverse coded.
Interpersonal Support Evaluation List (ISEL) | Baseline, 12 and 24 weeks
  This is a 12-item measure that assesses the perceived availability of social support from family, friends, and others. Each statement is scored using a 4-point scale (definitely false, probably false, probably true, definitely true) to measure subscales of appraisal, belonging, and tangible support. All items are summed to a total score ranging from 0 to 36 with higher scores indicating greater perceived social support.
Patient Health Questionnaire (PHQ-9) | Baseline, 12 and 24 weeks
  The PHQ-9 is a 9-item self-report measure that assesses the frequency of symptoms of major depressive disorder. Response options range from 0 ("not at all") to 3 (nearly every day). Total scores on the PHQ-9 range from 0-27 with greater scores indicating greater frequency of depressive symptoms.
Generalized Anxiety Disorder 7 (GAD-7) | Baseline, 12 and 24 weeks
  The 7-item GAD-7 will measure symptoms of anxiety. Items are scored 0-3, resulting in a total score of 0-21. Higher scores indicate more symptoms of anxiety.
Short Form Survey (SF-12) | Baseline, 12 and 24 weeks
  The SF-12 covers domains including: (1) physical functioning; (2) role-physical; (3) bodily pain; (4) general health; (5) vitality; (6) social functioning; (7) role emotional; and (8) mental health. Summary scores are calculated by summing factor-weighted scores across all 8 subscales, with factor weights derived from a US-based general population sample. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q-SF) | Baseline, 12 and 24 weeks
  Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-LES-Q-SF) consists of 14 items, assesses satisfaction with a variety of life domains such as physical health, work, and social relationships. The scoring of the Q-LES-Q-SF involves summing only the first 14 items to yield a raw total score. The last two items are not included in the total score but are standalone items. The raw total score ranges from 14 to 70. Higher level of enjoyment and satisfaction with life are reflected in higher scores.

OTHER OUTCOMES:
Percentage of eligible patients that agree to participate in the study | Approximately 15 months (recruitment study period)
  This will be done for acceptability with a target = 60%
Percentage of participants assigned to either intervention arm that complete any intervention session | 6 months
  The percentage of participants assigned to either intervention arm that complete any intervention session (target = 90%)
Percentage of participants assigned to either intervention arm that complete at least 3 of 4 sessions of the initially (first) assigned intervention | 3 months
  This will be done for acceptability with a target = 75%.
Percentage of participants that complete 3 of 4 sessions of the second intervention | 3 months
  This will be done for acceptability with a target = 50%.
Percentage of participants that complete any sessions of the second intervention | 3 months
  This will be done for acceptability with a target = 65%.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pfeiffer, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan (Michigan Medicine)-Brighton Health Center, Brighton, Michigan
  - University of Michigan (Michigan Medicine)-Canton Center, Canton, Michigan

IPD SHARING:
Plan to Share IPD: Yes
The Principal investigator (PI) will share information about this/these trial(s) via timely registration, updates, and results reporting in ClinicalTrials.gov in accordance with NIH policy.
  The PI will also upload data gathered in this proposal to an National Institute of Mental Health (NIMH)-designated central data, NIMH Data Archive (NDA), as prescribed by NOT-MH-15-012, working with NIMH program to determine the timing and extent of data sharing. This includes formulation of an enrollment strategy that will obtain the information necessary to generate a Global Unique Identifier (GUID) for each participant.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be entered into the NDA within 1 year of the conclusion of the study.
Access Criteria: No additional access restrictions will be placed on the de-identified data beyond those that are standard for the NDA.
URL: https://nda.nih.gov